CLINICAL TRIAL: NCT02146495
Title: Mechanistic Perspective on EEG Based Amygdala Driven NF in Fibromyalgia
Brief Title: Targeted Limbic Self-modulation as a Potential Treatment for Patients Suffering From Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TASMC-14-HS-0044-CTIL
Record Dates: First submitted 2014-05-21; First posted 2014-05-23 (Estimated); Last update posted 2024-03-20 (Actual); Status verified 2024-02

CONDITIONS: Fibromyalgia (FM)
Keywords: Fibromyalgia, neurofeedback, fMRI, EEG
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Simultaneous EEG/ fMRI Recordings during Amyg-EFP-NF (Experimental): Patients with FM will undergo concurrent EEG and fMRI recordings. During the fMRI scans, they will engage in Amyg-EFP NF training.
  Interventions: Device: Simultaneous EEG and fMRI recordings
- Amyg-EFP-NF Trial (Active Comparator): The EFP-NF procedure will include a multisession NF trial (10 sessions) using feedback driven by the Amyg-EFP model.
  Interventions: Device: Amygdala-Electrical Fingerprint (Amyg-EFP)-NF Trial
- Amyg-EFP-NF Sham Trial (Sham Comparator): The sham NF procedure will include a multisession NF trial (10 sessions) using sham feedback; in this condition, the feedback will be provided based on a randomized Amyg-EFP signal.
  Interventions: Device: Amygdala-Electrical Fingerprint (Amyg-EFP)-NF Sham Trial
- Treatment As Usual (No Intervention): Patients in this group will continue their usual treatment without any intervention. Patients in this control group will undergo a complete clinical and neural evaluation at the beginning and end of a defined period, similar to the NF intervention period, and a clinical follow-up (after 10-12 months).

INTERVENTIONS:
Device: Simultaneous EEG and fMRI recordings
  Arms: Simultaneous EEG/ fMRI Recordings during Amyg-EFP-NF
Device: Amygdala-Electrical Fingerprint (Amyg-EFP)-NF Trial — Neurofeedback training utilizing Amygdala Electrical Fingerprint (Amyg-EFP) methodology
  Arms: Amyg-EFP-NF Trial
Device: Amygdala-Electrical Fingerprint (Amyg-EFP)-NF Sham Trial — Sham neurofeedback training based on a randomized artificial Amyg-EFP signal.
  Arms: Amyg-EFP-NF Sham Trial

SUMMARY:
The goal of this study is to test whether voluntary regulation of limbic system activation is possible in patients with fibromyalgia and to examine the neurobehavioral effects of specific neuromodulation of this circuit on somatosensory, limbic, and cognitive processes. This goal will be achieved by using a method previously developed for the construction of an fMRI-enriched EEG model ("EEG-Finger-Print", EFP) that selectively targets the amygdala BOLD activation (Amyg-EFP). The investigators conducted two studies: In the first study, the investigators conducted simultaneous recordings of EEG and fMRI during Amyg-EFP NF training on patients with FM. The main objective is to demonstrate target engagement following Amyg-EFP-NF training in FM patients. In the second study, the investigators aim to conduct a randomized clinical trial to examine the causal effect of the Amyg-EFP NF trial. The investigators will compare neurobehavioral effects between three groups. I. Amyg-EFP-NF group: a multisession NF trial using the Amyg-EFP model. II. Control group 1- sham-NF: a multisession NF trial using sham feedback. III. Control group 2: patients in this group will continue their usual treatment without intervention.

DETAILED DESCRIPTION:
The current study aims to focus on the neural mechanism and brain-guided therapy of Fibromyalgia (FM); a chronic pain syndrome. Despite intense investigations, the pathophysiology of fibromyalgia remains elusive. Several studies demonstrated that morphological and functional changes in the central nervous system may play an important role in FM development and progression. The unknown etiopathology of FM contributed greatly to the absence of mechanism-specific cures. The insufficient treatment for FM, along with the understanding that CNS abnormality constitutes a major factor in FM pathophysiology, emphasizes the need for mechanism-based therapeutic intervention and opens the door for advanced neuromodulation techniques. Guided by this approach, the investigators aspired to establish a multi-function model with the potential to exert neuromodulation effects. To address this goal, the investigators employ a method previously developed for the construction of an fMRI-enriched EEG model ("EEG-Finger-Print", EFP). In this approach, EEG is used to predict specific brain activity, as measured by fMRI in a given region. Our main objective is to explore the neural mechanisms that underlie limbic neuromodulation and to gain a profound understanding of the functional processes that can potentially modify deficient functions in FM. The investigators intend to conduct two studies. In the first study, the investigators focus on the previously developed EFP model that selectively targets the amygdala BOLD activation (Amyg-EFP). The investigators aspired to investigate Amyg-EFP-NF effects on chronic pain in FM. To do so, the investigators conducted simultaneous recordings of EEG and fMRI during Amyg-EFP NF training on patients with FM. The main research objective of this study is to demonstrate target engagement following Amyg-EFP-NF training in FM patients. In the second study, the investigators aim to conduct a randomized clinical trial to examine the causal effect of the Amyg-EFP on patients with FM and to explore the clinical effect of this model on a wide range of symptoms related to FM. To examine the neural, clinical, and behavioral specific effects of the EFP-NF training, the investigators will implement a comprehensive clinical assessment. Furthermore, the investigators will conduct an MRI/fMRI scan before and after the EFP-NF trial, in order to explore the neural modification effects. Clinical follow-up will be conducted after 10-12 months from the post-intervention evaluation. The investigators will compare the neural, clinical, and behavioral effects between three groups. I. Amyg-EFP-NF group: a multisession NF trial using feedback driven by the Amyg-EFP model. II. Control group I- sham-NF: a multisession NF trial using sham feedback. III. Control group II: patients in this group will continue their usual treatment without any intervention. The investigators hypothesize that patients in the Amyg -EFP-NF group will exhibit wider and more robust changes in neural and behavioral outcomes associated with the wide range of symptoms related to FM. This study can significantly advance the understanding of the neural processes that mediate modification of somatic-affective functions in patients with FM and, therefore, enable the establishment of better treatment prediction and possibly more personalized procedures in future studies.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-55
* Fibromyalgia diagnosis by a specialist in internal medicine, Neurology or Pain medicine
* Subjective complaints about sleep disorder
* Pain does not stop despite regular medication- at least three events per week of pain ranked five out of ten
* chronic drug treatment should not be change in the near future (6 weeks).
* Hebrew speaker
* Accepted criteria for MRI scan for medical use will be followed, according to the procedures prescribed in the MRI institute of the Tel-Aviv Sourasky medical center.

Exclusion Criteria:

* Non-Hebrew speakers
* Diagnosis of another pain chronic syndrome or any significant medical illness.
* History of psychiatric or neurological diseases requiring hospitalization.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2022-08 (Actual); Study Completion 2022-08 (Actual)

PRIMARY OUTCOMES:
Clinical improvement using the Fibromyalgia Impact Questionnaire (FIQ) to evaluate FM symptoms | Immediately post-intervention relative to the baseline level
  Scoring from 0 (no impairment) to 80 (maximum), with subscales ranging up to 10 (maximum).
Clinical improvement using the Symptom Severity Score (SSS) | Immediately post-intervention relative to the baseline level
  Ranges from 0 to 12 (highest severity).
Clinical improvement using the Widespread Pain Index (WPI) | Immediately post-intervention relative to the baseline level
  Ranges from 0 to 19 (highest level of pain distribution).
Clinical improvement using the SF-36 Health Survey (SF-36) to evaluate daily impacts of FM | Immediately post-intervention relative to the baseline level
  Scores from 0 to 100 (higher scores indicate better health).
Clinical improvement using the Trait Anxiety Inventory (STAI-T) to evaluate the level of anxiety | Immediately post-intervention relative to the baseline level
  Ranges from 20 to 80 (highest anxiety level).
Clinical improvement using the Beck Depression Inventory (BDI) to evaluate the level of depression | Immediately post-intervention relative to the baseline level
  Ranges from 0 to 63 (highest depression level).
Long-term clinical improvement using the Fibromyalgia Impact Questionnaire (FIQ) to evaluate FM symptoms | Change in symptoms at 10-12 months relative to the baseline level (Follow-up measure vs. Baseline)
  Scoring from 0 (no impairment) to 80 (maximum), with subscales ranging up to 10 (maximum).
Long-term clinical improvement using the Symptom Severity Score (SSS) | Change in symptoms at 10-12 months relative to the baseline level (Follow-up measure vs. Baseline)
  Ranges from 0 to 12 (highest severity).
Long-term clinical improvement using the Widespread Pain Index (WPI) | Change in symptoms at 10-12 months relative to the baseline level (Follow-up measure vs. Baseline)
  Ranges from 0 to 19 (highest level of pain distribution).
Long-term clinical improvement using the SF-36 Health Survey (SF-36) to evaluate daily impacts of FM | Change in symptoms at 10-12 months relative to the baseline level (Follow-up measure vs. Baseline)
  Scores from 0 to 100 (higher scores indicate better health).
Long-term clinical improvement using the Trait Anxiety Inventory (STAI-T) to evaluate the level of anxiety | Change in symptoms at 10-12 months relative to the baseline level (Follow-up measure vs. Baseline)
  Ranges from 20 to 80 (highest anxiety level).
Long-term clinical improvement using the Beck Depression Inventory (BDI) to evaluate the level of depression | Change in symptoms at 10-12 months relative to the baseline level (Follow-up measure vs. Baseline)
  Ranges from 0 to 63 (highest depression level).

SECONDARY OUTCOMES:
Neural Prediction | Through study completion, an average of 2 year
  Simultaneous fMRI/EEG scan in order to identify whether the Amyg-EFP signal reliably predicts the amygdala BOLD activity

OTHER OUTCOMES:
Brain pattern Changes | Change in neural pattern immediately post-intervention relative to the baseline level (Post-intervention vs. Baseline)
  Measured via real-time fMRI; region of interest analysis in the amygdala; comparison between post vs pre scans: change in blood-oxygen-level-dependent (BOLD) response to regulate > baseline condition during NF task.
Amyg-EFP-NF regulation success | 1-10 weeks
  Measured by change in Amyg-EFP power; based on the difference between regulate and baseline conditions during the neurofeedback cycles
Pain Assessment | Change in pain level immediately post-intervention relative to the baseline level (Post-intervention vs. Baseline)
  Quantitative Sensory Testing (QST)- which assesses somatosensory function and provides thermal pain thresholds and sensory threshold.
Sleep assessment | Change in sleep quality immediately post-intervention relative to the baseline level (Post-intervention vs. Baseline)
  The investigators were measured via one-night sleep monitoring using the WatchPAT-200 device.
  While the specific range scores for sleep latency and sleep efficiency using the WatchPAT-200 are not explicitly detailed in the available documentation, it's generally accepted in sleep studies that normal sleep efficiency is considered to be 85% or higher. Normal sleep onset latency typically ranges from 10 to 25 minutes.
  To evaluate sleep quality, the investigators calculate a combined score using two sleep metrics: sleep latency and sleep efficiency.

CONTACTS AND LOCATIONS:
Overall Officials: Ayelet Or-Borichev, PhD, Principal Investigator — Sagol Brain Institute, Tel Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, N/A = Not Applicable, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Or-Borichev A, Lerner Y, Hamrani Y, Gurevitch G, Mor N, Doron M, Sarna N, Ablin JN, Hendler T, Sharon H. Targeted limbic self-neuromodulation for alleviating central sensitization symptoms in fibromyalgia. BMC Med. 2025 May 28;23(1):304. doi: 10.1186/s12916-025-04138-3. PMID 40437546